CLINICAL TRIAL: NCT02539381
Title: Stroke Vision: A Screening Tool for the Assessment of Visual Impairments in Stroke Survivors
Brief Title: The Stroke Vision App: A Screening Tool for Visual Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: GN15NE064
Record Dates: First submitted 2015-07-16; First posted 2015-09-03 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-08

CONDITIONS: Eye Abnormalities; Stroke
MeSH Terms: conditions — Eye Abnormalities; Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gold Standard Assessments (Other): * Formal perimetry (Goldman or Octopus visual field)
  * Albert's visual inattention test
  * Star cancellation visual inattention test
  * line bisection test
  * These are performed as part of the routine assessment in the visual stroke orthoptic clinic and neuro-ophthalmology clinics.
  * The time to perform the assessments or if the participant is unable to complete the assessment will be recorded.
  * Researcher will record a score (0-10) to quantify the participant's compliance
  Interventions: Procedure: Formal Perimetry (Goldman or Octopus visual Field); Procedure: Albert's visual inattention test; Procedure: Star cancellation visual inattention test
- Usual Clinical Screening Practice (Other): * Visual field assessment to confrontation
  * Visual inattention assessment to bilateral stimuli
  * The time to perform the assessments or if the participant is unable to complete the assessment will be recorded.
  * Researcher will record a score (0-10) to quantify the participant's compliance
  Interventions: Procedure: Visual field assessment to confrontation; Procedure: Visual inattention assessment to bilateral stimuli
- Stroke Vision App (Other): * Digital tumbling E visual accuity assessment
  * Digital visual field assessment
  * Digital line crossing assessment
  * Digital shape cancellation assessment
  * The time to perform the assessments or if the participant is unable to complete the assessment will be recorded.
  * Researcher will record a score (0-10) to quantify the participant's compliance
  Interventions: Device: Digital tumbling E visual accuity assessment; Device: Digital visual field assessment; Device: Digital line crossing assessment; Device: Digital shape cancellation assessment

INTERVENTIONS:
Procedure: Formal Perimetry (Goldman or Octopus visual Field)
  Arms: Gold Standard Assessments
Procedure: Albert's visual inattention test
  Arms: Gold Standard Assessments
Procedure: Star cancellation visual inattention test
  Arms: Gold Standard Assessments
Procedure: Visual field assessment to confrontation
  Arms: Usual Clinical Screening Practice
Procedure: Visual inattention assessment to bilateral stimuli
  Arms: Usual Clinical Screening Practice
Device: Digital tumbling E visual accuity assessment
  Arms: Stroke Vision App
Device: Digital visual field assessment
  Arms: Stroke Vision App
Device: Digital line crossing assessment
  Arms: Stroke Vision App
Device: Digital shape cancellation assessment
  Arms: Stroke Vision App

SUMMARY:
Visual impairment can affect up to 70% of stroke survivors, but many do not have their vision adequately assessed in hospital. An unidentified visual defect can cause significant problems for recovery and quality of life. The Stroke Vision app (an application currently scaled for a 10" Android tablet) has been developed to act as a screening tool for visual problems in stroke survivors; to help identify visual problems earlier and thereby improve rehabilitation outcomes. The app includes a suite of tests for assessing the patient's acuity, their visual fields and to aid in the identification of visual neglect / inattention. Furthermore, it includes educational information on visual stroke in order to better educate staff, patients and their carers. This study seeks to validate the novel digital assessments included in the Stroke Vision app against the current methods used for screening (clinical examination by confrontation field testing). Both screening measures will be compared with the gold standard methods for visual assessments, Octopus perimetry for fields and paper-based methods for visuospatial neglect

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to Visual Stroke Orthoptic Clinics
* All patients with stroke or stroke-like visual problems (for example, but not limited to bitemporal hemianopia caused by pituitary adenoma) referred to the neuro-ophthalmology clinics.
* Consent Provided

Exclusion Criteria:

* No spoken English
* Unable to provide consent
* Profound cortical blindness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Stroke Vision Tablet App to support assessment of visual field defects when compared with visual field assessment to confrontation in standard clinical practice | All assessments will be conducted following consent at standard clinical assessment visit
  Visual field will be captured either by the Stroke Vision App or by confrontation. Visual field will be reported by assessors (blinded to referral and comparator assessment) as either defect present, no defect present or unable to test. Agreement between visual field assessment supported by the Stroke Vision App and visual field assessment to confrontation in standard clincial practice will be quantified by the Kappa statistic. Accuracy metrics of sensitivity/specificity/predictive values will also be reported.
Accuracy of Stroke Vision Tablet App to support assessment of visual inattention defects when compared to visual inattention assessment to bilateral stimuli in standard clinical practice | All assessments will be conducted following consent at standard clinical assessment visit
  Visual inattention tests will be conducted either by the Stroke Vision App or by inattention to bilateral stimuli in standard clinical practice. Inattention will be reported by assessors (blinded to referral and comparator assessment) as either defect present, no defect present or unable to test. Agreement between visual inattention assessment supported by the Stroke Vision App and inattention to bilateral stimuli in standard clincial practice will be quantified by the Kappa statistic. Accuracy metrics of sensitivity/specificity/predictive values will also be reported.

SECONDARY OUTCOMES:
Accuracy of Stroke Vision Tablet App to support assessment of visual field defects when compared with "Gold standard" formal perimetry assessments | All assessments will be conducted following consent at standard clinical assessment visit
  Visual field will be captured either by the Stroke Vision App or by formal perimetry assessments. Visual field will be reported by assessors (blinded to referral and comparator assessment) as either defect present, no defect present or unable to test. Agreement between visual field assessment supported by the Stroke Vision App and visual field assessment to formal perimetry will be quantified by the Kappa statistic. Accuracy metrics of sensitivity/specificity/predictive values will also be reported.
Accuracy of Stroke Vision Tablet App to support assessment of visual inattention defects when compared with "Gold standard" Albert's visual inattention test, Star cancellation visual inattention test, Line Bisection test | All assessments will be conducted following consent at standard clinical assessment visit
  Visual inattention tests will be conducted either by the Stroke Vision App or by Gold standard" Albert's visual inattention test, Star cancellation visual inattention test, Line Bisection test conducted by a clinician. Inattention will be reported by assessors (blinded to referral and comparator assessment) as either defect present, no defect present or unable to test. Agreement between visual inattention assessment supported by the Stroke Vision App and "Gold standard" Albert's visual inattention test, Star cancellation visual inattention test, Line Bisection test will be quantified by the Kappa statistic. Accuracy metrics of sensitivity/specificity/predictive values will also be reported.

OTHER OUTCOMES:
Proportion of patients completing Gold standard vision assessments | All assessments will be conducted following consent at standard clinical assessment visit
Proportion of patients competing usual clinical practice vision assessments | All assessments will be conducted following consent at standard clinical assessment visit
Proportion of patients competing Stroke vision app assessments | All assessments will be conducted following consent at standard clinical assessment visit
Time to complete Gold standard vision assessments | All assessments will be conducted following consent at standard clinical assessment visit
Time to complete usual clinical practice vision assessments | All assessments will be conducted following consent at standard clinical assessment visit
Time to complete Stroke vision app assessments | All assessments will be conducted following consent at standard clinical assessment visit

CONTACTS AND LOCATIONS:
Overall Officials: Christine McAlpine, MBChB FRCP, Principal Investigator — NHS Greater Glasgow & Clyde
Locations (1):
- Gartnavel General Hospital, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Derived] Quinn TJ, Livingstone I, Weir A, Shaw R, Breckenridge A, McAlpine C, Tarbert CM. Accuracy and Feasibility of an Android-Based Digital Assessment Tool for Post Stroke Visual Disorders-The StrokeVision App. Front Neurol. 2018 Mar 28;9:146. doi: 10.3389/fneur.2018.00146. eCollection 2018. PMID 29643830